CLINICAL TRIAL: NCT00879905
Title: A Phase I Dose Escalation, Multi-center, Open-label Study of HSP990 Administered Orally in Adult Patients With Advanced Solid Malignancies
Brief Title: A Study of HSP990 Administered by Mouth in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHSP990A2101; 2008-006440-19 (EudraCT Number)
Record Dates: First submitted 2009-04-09; First posted 2009-04-13 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2012-10

CONDITIONS: Advanced Solid Malignancies
Keywords: Phase I; Adults; HSP990; Advanced Solid Tumors; Hsp90 inhibitor; Cancer
MeSH Terms: conditions — Neoplasms | interventions — 2-amino-7-(4-fluoro-2-(6-methoxypyridin-2-yl)phenyl)-4-methyl-7,8-dihydropyrido(4,3-d)pyrimidin-5(6H)-one

ARMS (2):
- once weekly dosing schedule (Experimental)
  Interventions: Drug: HSP990
- twice weekly dosing schedule (Experimental)
  Interventions: Drug: HSP990

INTERVENTIONS:
Drug: HSP990

SUMMARY:
This study will study the safety, tolerability and metabolism of a drug called HSP990 when given by mouth once a week or twice weekly to subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed, advanced malignant solid tumors whose disease has progressed on standard therapy or for whom no standard therapy exists
2. All patients must have at least one measurable lesion as defined by RECIST. Irradiated lesions are only evaluable for disease progression
3. All patients must have documented progressive disease before entering the study
4. Age ≥ 18 years
5. World Health Organization (WHO) Performance Status ≤ 2
6. Life expectancy of ≥ 12 weeks
7. Patients must have the certain laboratory values
8. Patients able and willing to swallow capsules
9. Ability to understand the patient information and informed consent form and comply with the protocol
10. Signed and dated written informed consent is available
11. Only for patients enrolled at MTD: willing to provide a fresh pre-dose and post-dose tumor biopsy.

Exclusion Criteria:

1. Patients with present or history of CNS metastasis.
2. Prior treatment with any Hsp90 or HDAC inhibitor compound.
3. Patients who have not recovered from side effects of previous systemic anticancer therapy to < CTCAE Grade 2 prior to the first dose
4. Patients identified to be "poor or intermediate CYP2C9 metabolizers"
5. Patients who received systemic anti-cancer treatment prior to the first dose of HSP990 within the following time frames:

   * Patients who have received cyclical chemotherapy within a period of time that is shorter than the cycle length used for that treatment (e.g., 6 weeks for nitrosourea, mitomycin-C) prior to starting study drug or who have not recovered from the side effects of such therapy
   * Patients who have received biologic therapy (e.g., antibodies) within a period of time that is ≤ 4 weeks prior to starting study drug or who have not recovered from the side effects of such therapy
   * Patients who have been treated with a continuous or intermittent small molecule therapeutic within a period of time that is ≤ 5 t1/2 or ≤ 4 weeks (whichever is shorter) prior to starting study drug or who have not recovered from the side effects of such therapy
   * Patients who have received any other investigational agents within a period of time that is ≤ 5 t1/2 or less than the cycle length used for that treatment or ≤ 4 weeks (whichever is shorter) prior to starting study drug or who have not recovered from the side effects of such therapy
   * Patients who have received wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
   * Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
6. Treatment with therapeutic doses of sodium warfarin (Coumadin).
7. Patients using medications that are CYP2C9 inhibitors and/or medications known to have QT prolongation effect and cannot be switched or discontinued to an alternative drug prior to commencing HSP990 dosing.
8. Unresolved diarrhea ≥ CTCAE grade 2
9. Patients who do not have either an archival tumor sample available or readily obtainable in the course of the study or are unwilling to have a fresh tumor sample collected at baseline.
10. Pregnant or lactating women.
11. Fertile women of childbearing potential (WCBP) not using adequate contraception (abstinence, oral contraceptives, intrauterine device or barrier method of contraception in conjunction with spermicidal jelly or surgically sterile). Male patients whose partners are WCBP, not using adequate contraception.
12. Acute or chronic liver disease.
13. Acute or chronic renal disease.
14. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of HSP990
15. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol.
16. Known diagnosis of HIV infection (HIV testing is not mandatory).
17. Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
18. Cardiac exclusion criteria:

    * History (or family history) of long QT syndrome.
    * Mean QTcF ≥ 480 msec on screening ECG
    * History of clinically manifest ischemic heart disease including myocardial infarction, or unstable angina ≤ 3 months prior to study start.
    * Left ventricular (LV) dysfunction (LVEF ≤ 45%) by MUGA or ECHO
    * Clinically significant ECG abnormalities including one or more of the following: left bundle branch block (LBBB), right bundle branch block (RBBB) with left anterior hemiblock (LAHB), or 3rd degree AV block.
    * History or presence of atrial fibrillation, atrial flutter or ventricular arrhythmias including ventricular tachycardia or Torsades de Pointes.
    * Clinically significant resting bradycardia (< 50 beats per minute).
    * Patients who are currently receiving treatment with any medication which has a relative risk or prolonging the QTcF interval or inducing Torsades de Pointes (as listed in Post-text supplement 2) and cannot be switched or discontinued to an alternative drug prior to commencing HSP990 dosing.
    * Obligate use of a cardiac pacemaker.
    * Other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of HSP990 in patients treated once weekly or twice weekly | At the end of the dose escalation phase of the study

SECONDARY OUTCOMES:
True DLT rate | At the end of the 1st 4 weeks of treatment
Preliminary Efficacy | Every 2 months (or 8 weeks, which equals 2 treatment cycles)
Drug metabolism in Humans, PK, PD | every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Toronto, Ontario, Canada
- Novartis Investigative Site, Toulouse, France
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- See also: Results for CHSP990A2101 can be found on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9063